CLINICAL TRIAL: NCT04180150
Title: A Randomized, Double-blinded, Placebo-controlled, Phase IIa Study of TQ-A3334 Combined With Entecavir in the Treatment of Untreated or HBV DNA Negative Subjects With Chronic Hepatitis B
Brief Title: A Study of TQ-A3334 Combined With Entecavir in the Treatment of Chronic Hepatitis B
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TQ-A3334-II-01a
Record Dates: First submitted 2019-11-26; First posted 2019-11-27 (Actual); Last update posted 2019-12-16 (Actual); Status verified 2019-10

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQ-A3334 combined with entecavir (Experimental): Subjects receive TQ-A3334 (1.2 mg QW) and entecavir (0.5 mg qd) in 24 weeks
  Interventions: Drug: TQ-A3334; Drug: Entecavir Tablet
- Placebo combined with entecavir (Placebo Comparator): Subjects receive placebo (0 mg QW) and entecavir (0.5 mg qd) in 24 weeks
  Interventions: Drug: Placebo; Drug: Entecavir Tablet

INTERVENTIONS:
Drug: TQ-A3334 — TQ-A3334 is a kind of TLR7 receptor agonist.
  Arms: TQ-A3334 combined with entecavir
Drug: Placebo — Placebo is a treatment which is designed to have no therapeutic value.
  Arms: Placebo combined with entecavir
Drug: Entecavir Tablet — Entecavir (ETV) tablet is an antiviral medication used in the treatment of hepatitis B virus (HBV) infection.

SUMMARY:
This is a randomized, double-blinded, placebo-controlled, phase IIa study to evaluate safety and efficacy of TQ-A3334 combined with entecavir in the untreated or HBV DNA negative subjects with Chronic Hepatitis B.

ELIGIBILITY:
Inclusion Criteria:

* 1. 18 and 65 years old ; 2. HBsAg positive at least for 6 months ; 3. HBeAg positive chronic hepatitis B, HBV DNA > 10^5 copies/ml; 4. Fibroscan ≤ 12.4 Kpa，2×ULN ≤ ALT ≤ ULN; 5. New diagnosed chronic hepatitis B subjects;

Exclusion Criteria:

* 1.Combined with other virus infection ; 2.Has cirrhosis or hepatocellular carcinoma; 3.Has autoimmune diseases; 4.Has thyroid disease; 5.Has eye diseases; 6.Has clinically significant abnormalities/diseases ≥ grade 2; 7.Has history of chronic kidney disease, renal insufficiency, renal anemia; 8.Peripheral blood index is low; 9.Has a history of allergy to experimental drugs or their excipients; 10.Has participated in other clinical trials within 3 months; 11.Breastfeeding or pregnant women.; Men unwilling to use adequate contraceptive measures during the study; 12.According to the judgement of the researchers, there are other factors that subjects are not suitable for the study.; 13.Has history of drug abuse in the past five years;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Cmax | Hour 0, 5, 10, 20, 30 minutes, 1, 2 , 3 , 6 , 12, 24, 72 , 168 hours post-dose at week 1 and week 12; Hour 0 of week 4, week 7, week 9, week 11.
  Cmax is the maximum plasma concentration of TQ-A3334 or metabolite(s).
Tmax | Hour 0, 5, 10, 20, 30 minutes, 1, 2 , 3 , 6 , 12, 24, 72 , 168 hours post-dose at week 1 and week 12; Hour 0 of week 4, week 7, week 9, week 11.
  To characterize the pharmacokinetics of TQ-A3334 by assessment of time to reach maximum plasma concentration.
AUC0-t | Hour 0, 5, 10, 20, 30 minutes, 1, 2 , 3 , 6 , 12, 24, 72 , 168 hours post-dose at week 1 and week 12; Hour 0 of week 4, week 7, week 9, week 11.
  To characterize the pharmacokinetics of TQB3804 by assessment of area under the plasma concentration time curve from zero to infinity.
Cytokine | Hour 0, 1.5 , 12 , 24 , 72 hours post-dose at week 1 and week 12; Hour 0 at week 7.
  Including IFN-α, IFN-γ, TNF-α, IL-6, IL-2, MCP-1 and so on.

SECONDARY OUTCOMES:
HBV biomarker | Day 1 pre-dose, day 84, day 168, day 336 post-dose.
  Including HBsAg, HBsAb, HBeAb, anti-HBc, HBV-DNA, HBV RNA and HBcrAg.
Lymphocyte function | Hour 0 pre-dose, day 56, day 84, day 168 at post-dose.
  Analysis of immune cell response to hepatitis B antigen after treatment.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The second affiliated hospital of chongqing medical university, Chongqing, Chongqing Municipality
  - The first hospital of Jilin University, Changchun, Jinlin